CLINICAL TRIAL: NCT00207974
Title: Pharmacokinetic Study of Marine Active in Health Men
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: China Medical University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMR94-IRB-68
Record Dates: First submitted 2005-09-16; First posted 2005-09-21 (Estimated); Last update posted 2005-11-17 (Estimated); Status verified 2005-09

CONDITIONS: Hyperuricemia, Anserine, Pharmacokinetic
Keywords: Hyperuricemia, Anserine, Pharmacokinetic
MeSH Terms: conditions — Hyperuricemia

INTERVENTIONS:
Drug: Marine active

SUMMARY:
Hyperuricemia is often associated with metabolic syndrome, which is a known precursor of atherosclerosis. The Yaizu Suisankagaku Industry Company have developed industrial production, named Marine Active. Human clinical trials showed reduction of creatine phosphokinase activity and sero-uric acid. Randomize, double blind clinical trial is entrust to our hospital. This study design is blood sampling from the health men who take 1 gm of marine active to analyse the pharmacokinetics of anserine.

DETAILED DESCRIPTION:
Hyperuricemia is a common metabolic disorder. It can result from a decreased renal uric acid excretion, increased urate production, or both. The classical association with clinical gout is well-known. The principal indications for uric acid-lowering therapy, including allopurinol, probenecid and sulfinpyrazone, are the patients with gout history, macroscopic subcutaneous tophi, frequent attacks of gouty arthritis, or a documented state of uric acid overproduction. Hyperuricemia is often associated with metabolic syndrome,which is known a percursor of atherosclerosis. For the gout attack only 5% per year of the hyperuricemic population, medical management is not indicated for patients without gouty arthritis. Diet control is the leading way to control serum uric acid level, but usually it is not enough. So how to management hyperuricemia is important and is a potential management.Histidine-containing dipeptides such as Anserine and Carnosine have been studied extensively in recent years. These dipeptides were shown to be effective in acting as buffering agents against protons developed during anaerobic exercise. Anserine and Carnosine also have strong anti-oxidant activity, anti-cancer activity, immuno-response modulation, fat reduction and enhanced wound healing functions. The Yaizu Suisankagaku Industry Company have developed industrial production process to extract and purify the dipeptides from Bonito and Tuna. The extract, named Marine Active, was able to offer anti-fatigue activity by animal trial data. Human clinical trials showed reduction of creatine phosphokinase activity and sero-uric acid. Randomize, double blind clinical trial is entrust to our hospital. This study design is blood sampling from the health men who take 1 gm of marine active to analyse the pharmacokinetics of anserine.

ELIGIBILITY:
Inclusion Criteria:

-Male volunteers, age between 20 to 35 years

Exclusion Criteria:

* Chronic medical history
* Significant liver or renal dysfunction,
* Have been administrated by any drug within 2 weeks before the initiation of study.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Chin Huang, MD, Principal Investigator — Chinese-Western Medicine Cooperation, China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan